CLINICAL TRIAL: NCT05188430
Title: A Double-blind, Randomized, Placebo-controlled Clinical Trial on the Metabolic Effect of an Innovative Chitosan Formulation
Brief Title: Metabolic Effect of an Innovative Chitosan Formulation
Acronym: CHITOCHOL
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Bologna (Other)
Responsible Party: Principal Investigator, Arrigo F.G. Cicero, Professor, University of Bologna
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Chito_RCT2022
Record Dates: First submitted 2021-12-09; First posted 2022-01-12 (Actual); Last update posted 2022-01-12 (Actual); Status verified 2021-12

CONDITIONS: Hypercholesterolemia; Overweight and Obesity
Keywords: Hypercholesterolemia; Overweight; Class I obesity; Low-density lipoprotein cholesterol; Lipids; Chitosan; Medical device
MeSH Terms: conditions — Hypercholesterolemia; Overweight; Obesity | interventions — Equipment and Supplies

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active treatment (Active Comparator): Medical Device (Kaptufat®)
  Interventions: Device: Medical Device (Kaptufat®)
- Placebo (Placebo Comparator): Placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Device: Medical Device (Kaptufat®) — 140 mg chitosan, 460 mg cellulose and 35.384 mg ascorbic acid for 1 tablet
  Oral administration: 3 tablets twice a day before the main meals
  Arms: Active treatment
Other: Placebo — Oral administration: 3 tablets twice a day before the main meals
  Arms: Placebo

SUMMARY:
Chitosan is a natural polysaccharide of β-1,4-linked glucosamine residues deriving from chitin, a dietary fiber primarily obtained from fungal cell walls and the exoskeletons of various crustaceans (e.g. crab, lobster, and shrimp) and whose cholesterol-lowering properties are due to the hydrophobic bonds it forms with cholesterol and other sterols, interfering with the emulsification process in the intestine.

In addition to reducing low-density lipoprotein cholesterol (LDL-C) levels, several studies showed that chitosan administration may help reduce body weight. For this reason, its use might be particularly useful as a strategy to simultaneously control two different risk factors for the development of CVDs.

ELIGIBILITY:
Inclusion Criteria:

* Subjects agree to participate in the study and having dated and signed the informed consent form;
* Subjects who have the capability to communicate, to make themselves understood, and to comply with the study's requirements;
* Male or female aged ≥ 18 years and ≤ 70 years old;
* Subjects free from cardiovascular diseases (CVDs) (primary prevention for CVDs);
* Subjects with sub-optimal serum levels of cholesterol (total cholesterol (TC) of 200-240 mg/dl OR LDL-C of 130-190 mg/dl);
* Subjects with body mass index (BMI) 25 -34.9 Kg/m2

Exclusion Criteria:

* Subjects already affected by CVDs (secondary prevention for CVDs);
* Subjects with serum levels of triglycerides (TG)> 400 mg/dl;
* Type 1 or type 2 diabetes;
* Lipid-lowering treatment not stabilized since at least 2 months;
* Known current gastrointestinal diseases and use of medications for their treatment;
* Known clinically relevant decline in renal function;
* Women in fertile age not using consolidated contraceptive methods
* Pregnancy and Breastfeeding;
* History or clinical evidence of any significant concomitant disease that could compromise the safety of the subject or the possibility of completing the study;
* Any medical or surgical condition that would limit the patient adhesion to the study protocol

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-03-01 (Estimated); Primary Completion 2022-09-03 (Estimated); Study Completion 2022-09-03 (Estimated)

PRIMARY OUTCOMES:
Absolute change in LDL-C from baseline and between groups | 12 weeks
  Absolute change in LDL-C after 12 weeks of treatment with MD compared to placebo

SECONDARY OUTCOMES:
Absolute change in LDL-C from baseline and between groups | 6 weeks
  Absolute change in LDL-C from baseline and between groups after 6 weeks of treatment with MD compared to placebo
Absolute change in serum lipids other than LDL-C (TC, TG, HDL-C, non-HDL-C) and apolipoproteins from baseline and between groups | 12 weeks
  Absolute change in serum lipids other than LDL-C (TC, TG, HDL-C, non-HDL-C) and apolipoproteins from baseline and between groups after 12 weeks of treatment with MD compared to placebo
Absolute change in serum lipids other than LDL-C (TC, TG, HDL-C, non-HDL-C) and apolipoproteins from baseline and between groups | 6 weeks
  Absolute change in serum lipids other than LDL-C (TC, TG, HDL-C, non-HDL-C) and apolipoproteins from baseline and between groups after 6 weeks of treatment with MD compared to placebo
Absolute change in lipids ratios from baseline and between groups | 6 weeks
  Absolute change in lipids ratios from baseline and between groups after 6 weeks of treatment with MD compared to placebo
Absolute change in lipid accumulation product (LAP) from baseline and between groups | 6 weeks
  Absolute change in LAP from baseline and between groups after 6 weeks of treatment with MD compared to placebo
Absolute change in lipids ratios from baseline and between groups | 12 weeks
  Absolute change in lipids ratios from baseline and between groups after 12 weeks of treatment with MD compared to placebo
Absolute change in LAP from baseline and between groups | 12 weeks
  Absolute change in LAP from baseline and between groups after 12 weeks of treatment with MD compared to placebo
Absolute change in fasting plasma glucose (FPG) from baseline and between groups | 12 weeks
  Absolute change in FPG from baseline and between groups after 12 weeks of treatment with MD compared to placebo
Absolute change in fasting plasma insulin from baseline and between groups | 12 weeks
  Absolute change in fasting plasma insulin from baseline and between groups after 12 weeks of treatment with MD compared to placebo
Absolute change in fasting plasma glucose (FPG) from baseline and between groups | 6 weeks
  Absolute change in FPG from baseline and between groups after 6 weeks of treatment with MD compared to placebo
Absolute change in fasting insulin from baseline and between groups | 6 weeks
  Absolute change in fasting insulin from baseline and between groups after 6 weeks of treatment with MD compared to placebo
Absolute change in homeostatic model assessment for insuline resistance (HOMA-IR) index from baseline and between groups | 6 weeks
  Absolute change in HOMA-IR index from baseline and between groups after 6 weeks of treatment with MD compared to placebo
Absolute change in HOMA-IR index from baseline and between groups | 12 weeks
  Absolute change in HOMA-IR index from baseline and between groups after 12 weeks of treatment with MD compared to placebo
Absolute change in weight from baseline and between groups | 12 weeks
  Absolute change in weight from baseline and between groups after 12 weeks of treatment with MD compared to placebo
Absolute change in weight from baseline and between groups | 6 weeks
  Absolute change in weight from baseline and between groups after 6 weeks of treatment with MD compared to placebo
Absolute change in waist circumference from baseline and between groups | 6 weeks
  Absolute change in waist circumference from baseline and between groups after 6 weeks of treatment with MD compared to placebo
Absolute change in waist circumference from baseline and between groups | 12 weeks
  Absolute change in waist circumference from baseline and between groups after 12 weeks of treatment with MD compared to placebo
Absolute change in body mass index (BMI) from baseline and between groups | 12 weeks
  Absolute change in BMI from baseline and between groups after 12 weeks of treatment with MD compared to placebo
Absolute change in body mass index (BMI) from baseline and between groups | 6 weeks
  Absolute change in BMI from baseline and between groups after 6 weeks of treatment with MD compared to placebo
Absolute change in index of visceral adiposity index (VAI) from baseline and between groups | 6 weeks
  Absolute change in VAI from baseline and between groups after 6 weeks of treatment with MD compared to placebo
Absolute change in index of central obesity (ICO) from baseline and between groups | 6 weeks
  Absolute change in ICO from baseline and between groups after 6 weeks of treatment with MD compared to placebo
Absolute change in index of central obesity (ICO) from baseline and between groups | 12 weeks
  Absolute change in ICO from baseline and between groups after 12 weeks of treatment with MD compared to placebo
Absolute change in index of visceral adiposity index (VAI) from baseline and between groups | 12 weeks
  Absolute change in VAI from baseline and between groups after 12 weeks of treatment with MD compared to placebo

CONTACTS AND LOCATIONS:
Overall Officials: Arrigo F.G. Cicero, MD, PhD, Principal Investigator — AOU Policlinico S. Orsola-Malpighi
Locations (1):
- AOU Policlinico S.Orsola-Malpighi, Bologna, Italy